CLINICAL TRIAL: NCT07027046
Title: Application of da Vinci SP for Endometrial Cancer Surgical Staging: a Prospective Multicenter Study
Brief Title: Application of da Vinci SP for Endometrial Cancer Surgical Staging
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: SP endometrial cancer
Record Dates: First submitted 2025-05-30; First posted 2025-06-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Da Vinci SP Surgical Staging Group: Patients with early-stage endometrial cancer undergoing robotic surgical staging using the Da Vinci SP system.
  Interventions: Procedure: Robotic surgical staging

INTERVENTIONS:
Procedure: Robotic surgical staging — The intervention includes hysterectomy, bilateral salpingo-oophorectomy, and sentinel lymph node mapping, with possible lymphadenectomy or omentectomy, depending on histology.

SUMMARY:
Prospective Multicenter Observational Study The study involves the consecutive inclusion of every patient with endometrial cancer undergoing staging surgical treatment using a robotic approach with the da Vinci SP platform.

DETAILED DESCRIPTION:
The standard treatment for early-stage endometrial cancer is surgical staging, which includes total hysterectomy with bilateral salpingo-oophorectomy and surgical lymph node assessment.

The well-known advancements in minimally invasive surgery (MIS) have enabled laparoscopic and robotic surgical staging in gynecologic oncology. In the case of endometrial cancer, MIS is indeed the preferred surgical approach. Following the approval of the da Vinci Surgical System (Intuitive Surgical, Sunnyvale, CA, USA) for gynecological procedures by the United States Food and Drug Administration in 2005, the use of robotic surgery for endometrial cancer has significantly increased, with favorable outcomes even compared to conventional laparoscopy.

The growing need for increasingly less invasive surgical options has led to the development of the possibility to perform endometrial cancer surgical staging through a single abdominal incision. Despite several attempts to apply single-incision techniques to laparoscopy in the context of endometrial cancer, the standard minimally invasive approach for hysterectomy remains the four-trocar laparoscopic technique. One of the main reasons is that introducing both the endoscope and instruments through a single incision creates internal and external conflicts between instruments and the surgeon's hands. The parallel placement of surgical instruments leads to clashes and restricts the range of motion.

To overcome these limitations, robotic technology may be applied to the single-incision technique. The recent introduction of single-port robotic surgery with the fourth-generation da Vinci® SP Surgical System represents a technological advancement. In fact, the system's flexible articulation of instruments allows for more effective manipulation while reducing instrument collisions. Moreover, the flexible camera provides a new operational angle in all directions.

The new da Vinci SP Surgical System (SP) received regulatory approval for use in gynecologic surgery in Italy in 2024. However, to date, studies in the literature on the use of the da Vinci SP robot in patients with endometrial cancer are limited due to the relatively small number of patients, single-center settings, and the retrospective nature of most studies.

Because of these limitations in the literature, definitive evidence is still lacking regarding the efficacy and safety profile of the da Vinci SP in surgical staging of early-stage endometrial cancer.

Based on these premises, the aim of this study is to clarify the outcomes associated with this minimally invasive robotic approach by reporting one of the first experiences of robotic surgical staging for endometrial cancer using the new da Vinci SP robotic platform.

The primary objective of the study is to evaluate the surgical efficacy profile of the minimally invasive robotic approach using the da Vinci SP platform for the surgical staging of endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed endometrial carcinoma (including uterine carcinosarcoma)
* Performance status (ECOG) 0 - 1
* Patients undergoing staging surgery for endometrial cancer, including but not limited to robotic hysterectomy with bilateral salpingo-oophorectomy (ovarian preservation in selected patients is not an exclusion criterion) and possible sentinel lymph node biopsy/pelvic ± para-aortic lymphadenectomy
* Signed informed consent to participate in the study

Exclusion Criteria:

* Patients scheduled for an additional extra-genital surgical procedure during the staging surgery for endometrial carcinoma
* Patients with anesthesiological contraindications to a minimally invasive approach
* Synchronous tumor
* Recurrence of endometrial carcinoma
* Dementia or significantly altered mental status that may impair understanding and the ability to provide informed consent
* Any reason that may interfere with regular follow-up, even if limited to the first 30 days post-surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with histologically confirmed endometrial carcinoma at first diagnosis who have planned staging surgery for endometrial cancer to be performed using the robotic approach with the da Vinci SP platform
Sampling Method: Non-Probability Sample
Enrollment: 564 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Rate of satisfactory completion of staging surgery according to the criteria of national and international guidelines for the treatment of endometrial carcinoma. | 12 months
Rate of intraoperative complications, after categorization based on the type of complication and the timing of its occurrence. | 12 months
Rate of postoperative complications, after categorization based on the type of complication (within 30 days after surgery, after 30 days post-surgery) and according to the Clavien-Dindo classification. | 48 months

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) calculated from the date of randomization to the date of death from any cause or censored at the date of the last follow-up, after categorization based on molecular class and tumor prognostic factors. | up to 48 months (4 years)
Overall Survival (OS) calculated from the date of randomization to the date of death from any cause or censored at the date of the last follow-up, after categorization based on molecular class and tumor prognostic factors. | up to 48 months (4 years)
Quality of Life (QoL) assessed using the questionnaires from the EORTC QLQ-C30 (Version 3). | From baseline (pre-treatment) up to 48 months (4 years) post-randomization, with assessments every 6 months
Quality of Life (QoL) assessed using the questionnaires from EORTC QLQ-OV28. | From baseline (pre-treatment) up to 48 months (4 years) post-randomization, with assessments every 6 months
Quality of Life (QoL) assessed using the questionnaires from the EQ-5D-3L. | From baseline (pre-treatment) up to 48 months (4 years) post-randomization, with assessments every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vito Chiantera, MD, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (3):
- Italy (3):
  - Istituto Nazionale Tumori | "Fondazione Pascale", Napoli, Napoli
  - IEO - Istituto Europeo di Oncologia, Milan
  - Istituti Fisioterapici Ospitalieri - IFO, Roma